CLINICAL TRIAL: NCT01202006
Title: A Combined Diagnostic-therapeutic Strategy to Optimize Management of Patients With Previously Unrecognized Heart Failure in Primary Care
Brief Title: Strategy to Recognize and Initiate Treatment of Chronic Heart Failure
Acronym: STRETCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, F.H. Rutten, Dr. F.H. Rutten, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL31024.041.10
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Diagnosis; Treatment; Primary care
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): General practitioners of patients in the intervention group will receive detailed instructions on uptitration of ACE-inhibitors and beta-blockers before the inclusion of participants.
  Interventions: Other: Training of general practitioners in an uptitration protocol.
- Control (No Intervention): Patients in the control group receive care-as-usual. Their general practitioner will not be trained in applying the uptitration protocol.

INTERVENTIONS:
Other: Training of general practitioners in an uptitration protocol. — The general practitioners randomly allocated to the intervention group will be trained in the practical appliance of the Dutch GP's 'heart failure' guideline. They will receive detailed instructions on initiating diuretics with ACE-inhibitors and uptitration of ACE-inhibitors and beta-blockers.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a structured diagnostic-therapeutic strategy to detect and treat previously unrecognized (or unestablished) heart failure in primary care will improve the functional capacity, quality of care, the quality of life, and eventually the prognosis of these patients.

DETAILED DESCRIPTION:
Heart failure is an emerging epidemic in especially the elderly, with high mortality rates, substantial loss in quality of life, and high healthcare costs, mainly due to hospitalizations. The majority of (usually elderly) patients with heart failure are diagnosed and managed in primary care. However underdiagnosis and undertreatment of patients with heart failure in primary care are common. Implementation of a standardized diagnostic protocol together with educating general practitioners in a pragmatic treatment strategy in which the focus lays on uptitration of heartfailure medication, would fill the gap of underdiagnosis and undertreatment that nowadays exists in primary care.

All participants will undergo a standardized diagnostic work-up to establish or rule out heart failure. In those participants with an abnormal ECG and/or elevated natriuretic peptide level additional echocardiography will be performed at the outpatient clinic of the Diakonessenhuis in Zeist. The definite diagnosis of heart failure ('systolic' or 'diastolic') will be established by an expert panel consisting of two cardiologists and a general practitioner. The panel will apply the criteria of the updated heart failure guidelines (2008) of the European Society of Cardiology (ESC). Patients with heart failure will subsequently be treated by their own general practitioner. The participating general practitioners will be randomly divided into either care as usual (control group) or special uptitration (intervention group). Both groups will be using medication as recommended in the Dutch heart failure standard. However, general practitioners in the intervention group will be especially trained in the practical appliance of this guideline: the initiation of diuretics and ACE-inhibitors and structured uptitration of ACE-inhibitors and beta-blockers. In the training, practical examples will be used concerning barriers the general practitioners themselves encountered when using this medication. In the intervention group, patients with 'systolic' heart failure will receive the recommended maximal dose or the highest tolerated dose. Patients with 'diastolic' heart failure will receive optimal blood pressure and heart rate control with the preferred cardiovascular drugs. At baseline and six months after heart failure is established or ruled out, participants are asked to perform the six-minute walk test and fill out quality of life questionnaires. During those six months, only participants with heart failure will additionally fill out one of these questionnaires every three weeks. Also after six months, electronical files of the general practitioners will be scrutinized to assess the (dosage of) prescribed medication and visits to general practice and cardiology department.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or over
* Shortness of breath as reason for GP contact in the previous 12 months

Exclusion Criteria:

* Already established heart failure, that is a diagnosis of heart failure confirmed by the cardiologist with echocardiography
* A life expectancy shorter than 6 months
* Not being able to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 585 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of heart failure in elderly who presented to the general practitioner with shortness of breath on exertion. | one year
Differences in walking distance between the intervention and control group. | 6 months
  This outcome was added because of its relevance for patients with heart failure in April 2011. The change in study protocol was communicated to and approved by the Medical Ethics Committee of the UMC Utrecht.
Differences in quality of life between the intervention and control group. | 6 months
Differences in prescription of heart failure medication between the intervention and control group. | 6 months
Differences in (heart failure related) doctor-appointments and hospitalization rates between the intervention and control group. | 6 months

SECONDARY OUTCOMES:
Cost-effectiveness of the implemented diagnostic-therapeutic strategy. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frans H Rutten, MD, PhD, Principal Investigator — Julius Center for Health Sciences and Primary care
Locations (1):
- Julius Center for Health Sciences and Primary care, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] van Riet EE, Hoes AW, Limburg A, Landman MA, Kemperman H, Rutten FH. Extended prediction rule to optimise early detection of heart failure in older persons with non-acute shortness of breath: a cross-sectional study. BMJ Open. 2016 Feb 15;6(2):e008225. doi: 10.1136/bmjopen-2015-008225. PMID 26880668
- [Derived] van Riet EE, Hoes AW, Limburg A, van der Hoeven H, Landman MA, Rutten FH. Strategy to recognize and initiate treatment of chronic heart failure in primary care (STRETCH): a cluster randomized trial. BMC Cardiovasc Disord. 2014 Jan 8;14:1. doi: 10.1186/1471-2261-14-1. PMID 24400643